CLINICAL TRIAL: NCT06548633
Title: The Immediate Extent of the Hypoalgesic Effect Following Central Mobilisations to L3, L4 and L5
Acronym: HypoLumbar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Darren Cooper (Other)
Responsible Party: Sponsor-Investigator, Darren Cooper, Principal Lecturer in Sports Therapy, University of Worcester
Organization: University of Worcester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIEHEFCML345
Record Dates: First submitted 2024-08-02; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
Keywords: Vertebral Lumbar Mobilisations; Hypoalgesia; Pinprick sensitivity (PPS); Neuropen®
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The design of the study was a randomised, single-blind, repeated measures, cross-over design, performed in a single-centre environment.
Masking Description: The participants were blinded to the intervention they were receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vertebral Lumbar Mobilisations (Experimental): Participants received the intervention.
  Interventions: Other: Lumbar Vertebral Mobilisation

INTERVENTIONS:
Other: Lumbar Vertebral Mobilisation — The participants received Vertebral Lumbar Mobilisations, these were posterior-anterior central vertebral pressures (PACVPs) for four sets of 30 seconds, with up to 30s between each, at a grade III amplitude.

SUMMARY:
The aim of this study was to establish the efficacy of spinal mobilisations (a controlled application of a specific amount of force to a targeted spinal level) for reducing pain across different areas of the lower back. Pain was assessed using a pin prick sensation device and recorded in specific locations by the participant using a 10 cm line with one end indicating no pain and the other the worst pain possible.

DETAILED DESCRIPTION:
Study Design The design of the study was a randomised, single-blind, repeated measures, cross-over design, performed in a single-centre environment. Ethical approval was gained from the School of Sport and Exercise Science ethics committee at the University of Worcester (ISES2018RF1). Informed consent was gained from each participant before testing.

Sample and Inclusion Criteria The study included twenty asymptomatic participants (11 females and 9 males); the mean age of the participants was 21.9 years (±2.67, range 20- 30). A health questionnaire (based on the PARQ) was completed by each participant to establish any contraindications they may have to the experimental procedures, namely the application of vertebral mobilisations. No participants were required to be excluded as none of them had consulted their doctor in the last six months, were taking any medication, had an infection in the past two weeks, had no heart, asthma, diabetes, bronchitis, epilepsy or blood pressure issues, had any current muscle or joint injury, were able to train/exercise normally or knew of any other reason that would preclude them from participating.

Data Collection Each participant was randomly assigned using a random number generator to the order in which their lumbar vertebral levels were mobilised and to the order of each dermatome level tested for the baseline and all three mobilisation interventions.

Before initiating the experimental procedure, the participant's age, height, and weight were recorded. The participant was instructed to lay on their back, on the plinth and had the five locations for dermatome testing marked with a water-soluble pen. The researchers utilised the method of using participant's finger breadth to establish dermatome testing sites the dermatome testing sites were based on Keegan and Garrett's dermatome map. From this point forth, the spinal levels will be referred to as L2 or L3, respectively and the corresponding dermatome of the vertebral level will be referred to as DL2 or DL3.

Once these locations were marked on the participant's left leg, a demonstration of the Neuropen® (Owen Mumford, Oxfordshire, UK) was performed on the participant's hand (opposite to the side being tested). Once all this had been completed, baseline measures were taken. Using the Neuropen®, a standardised force of 40g was applied to one of the locations. The participant then received a small piece of card with a vertical 10cm visual analogue scale (VAS) line on it and a pen and was asked to draw a horizontal line on the scale to indicate how much sensation you feel, 0 being can-not feel anything and 10 being an extremely strong sensation. Following this explanation, the participant was asked if they understood and whether they needed further instruction to complete the VAS card. Once the participant marked the card, the card and pen were collected and stored, this process was repeated with the remaining four locations (these five cards provided the baseline data). A new tip was used for each participant, and a decrease in PPS represents a reduction in pain.

Once baseline measurements were collected by the lead researcher, the participant was asked to turn onto their front; the first (pre-determined) lumbar vertebra was found using the iliac crest as an anatomical landmark for the differentiation test. When the correct vertebra was located, the experimenter pressed record on the laptop connected to the PGD plinth to record the force applied and calculate the frequency.

The lumbar vertebra was mobilised using Maitland's vertebral mobilisation method for posterior-anterior central vertebral pressures (PACVPs) for four sets of 30 seconds with up to 30s between each, at a grade III amplitude and a target rate of 3Hz to ensure the total time for testing was less than fifteen minutes in duration, before the opioid system is activated. Once the fourth 30-second mobilisation had been completed, the researcher pressed stop on the laptop and asked the participant to roll onto their back. Then the next five sets of data were collected following the same procedure implemented for the baseline measures (collected in a different, pre-determined order each time). This process was repeated for the remaining two vertebrae.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and consent.

Exclusion Criteria:

* Yes to any Vertebral Mobilisation Contraindication.
* Consulted a doctor within the last 6 months?
* Presently taking any form of medication?
* Suffered from a bacterial or viral infection in the last 2 weeks?
* Ever suffered from any form of heart complaint?
* Family history of heart disease?
* Ever suffered from: Asthma, Diabetes, Bronchitis, Epilepsy, High blood pressure or Low blood pressure?
* Currently have any form of muscle or joint injury?
* Had to suspend training in the last two weeks for a physical reason?
* Is there anything that may prevent the successful completion of the tests that have been outlined?

Any "yes" answers to any of the questions above will require further detail, then the answers will be assessed to establish the potential risks to the participant and established if it is safe to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Pinprick sensitivity (PPS) | Up to 15 minutes
  Using a Neuropen® (Owen Mumford, Oxfordshire, UK) a standardised force of 40g was applied to one of the dermatome locations. The participant then received a small piece of card with a vertical 10cm visual analogue scale (VAS) line on it and a pen and was asked to "draw a horizontal line on the scale to indicate how much sensation you feel, 0 being can-not feel anything and 10 being an extremely strong sensation". Following this explanation, the participant was asked if they understood and whether they needed further instruction to complete the VAS card. Once the participant marked the card, the card and pen were collected and stored, this process was repeated with the remaining four locations (these five cards provided the baseline data). A new tip was used for each participant, and a decrease in PPS represents a reduction in pain.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Cooper, Dr, Study Director — University of Worcester
Locations (1):
- University of Worcester, Worcester, Worcestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be available upon request.
Supporting Information: Study Protocol, CSR
Time Frame: December 2024 onwards
Access Criteria: Emailing the study contact.
URL: https://www.worcester.ac.uk/about/profiles/dr-darren-cooper

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT06548633/Prot_SAP_000.pdf